CLINICAL TRIAL: NCT06941623
Title: Ultrasound Assessment for Comparison of Gastric Residual Volume After Ingestion of Carbohydrate Drink and Water in Obesity Class II and III Volunteers at Risk of Aspiration: A Randomized Crossover Study
Brief Title: Ultrasound Assessment for Comparison of Gastric Residual Volume After Ingestion of Carbohydrate Drink and Water in Obesity Class II and III Volunteers at Risk of Aspiration
Acronym: CarbDrinkUltra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Chanya Deekiatphaiboon, Anesthesiology department, Faculty of Medicine, Prince of Songkla University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: REC 66-538-8-1
Record Dates: First submitted 2024-03-08; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Gastroesophageal Reflux
Keywords: Carbohydrate drink; Gastric residual volume; Gastric ultrasound
MeSH Terms: conditions — Obesity; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate drink (Experimental): Volunteers receive a carbohydrate drink of 400 ml (50 g of glucose, clear color, same appearance, and containing bottles of water, prepared by the nutrition division, Songklanagarind hospital)
  Interventions: Diagnostic Test: Ultrasonography of gastric residual volume; Diagnostic Test: Point-of-care testing of glucose; Other: Hunger numeric rating scale; Other: Thirst numeric rating scale; Other: Nausea numeric rating scale
- Water (Placebo Comparator): Volunteers receive a bottle of 400 ml water (clear color, same appearance, and containing bottles of carbohydrate drink, prepared by the nutrition division, Songklanagarind hospital)
  Interventions: Diagnostic Test: Ultrasonography of gastric residual volume; Diagnostic Test: Point-of-care testing of glucose; Other: Hunger numeric rating scale; Other: Thirst numeric rating scale; Other: Nausea numeric rating scale

INTERVENTIONS:
Diagnostic Test: Ultrasonography of gastric residual volume — Gastric ultrasound will be performed by the radiologist on each participant before the study and at 0, 10, 20, 30, 60, 90, 120 minutes after drinking in the position of head upright 45 degree with left lateral decubitus to evaluate the gastric residual volume and time to empty gastric antrum. If time to empty gastric antrum is extended, ultrasound will be serial performed at 150 and 180 minutes.
  Other Names: GRV
Diagnostic Test: Point-of-care testing of glucose — We will perform the point-of-care test of glucose before the study and at 60, and 120 minutes after drinking.
  Other Names: POCT glucose, DTX
Other: Hunger numeric rating scale — Hunger will be measured by a numeric rating scale(NRS) before drinking, 60 and 120 minutes after drinking. The Numeric Rating Scale(NRS) is used for the self-report measurement of hunger levels, defined by numbers from 0 to 10, where 0 represents the lowest level of hunger and 10 represents the highest.
  Other Names: Hunger NRS
Other: Thirst numeric rating scale — Thirst will be measured by a numeric rating scale(NRS) before drinking, 60, and 120 minutes after drinking. The Numeric Rating Scale(NRS) is used for the self-report measurement of thirst levels, defined by numbers from 0 to 10, where 0 represents the lowest level of thirst and 10 represents the highest.
  Other Names: Thirst NRS
Other: Nausea numeric rating scale — Nausea will be measured by a numeric rating scale(NRS) before drinking, 60, and 120 minutes after drinking. The Numeric Rating Scale(NRS) is used for the self-report measurement of nausea levels, defined by numbers from 0 to 10, where 0 represents the lowest level of nausea and 10 represents the highest.
  Other Names: Nausea NRS

SUMMARY:
The goal of this clinical trial is to compare gastric residual volume between drinking a carbohydrate drink and water in obesity class II and III volunteers at risk of aspiration.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 35 kg/m2 (obesity class II and III)
* Gastroesophageal reflux disease and/or active gastroesophageal reflux symptoms in 6 months (heartburn and/or acid regurgitation)
* ASA status I-III
* NPO for 8 hours before the study

Exclusion Criteria:

* Chronic kidney disease or End-stage renal disease
* Diabetes Mellitus
* Use of any medication that affects gastric secretion or emptying within the past 24-hour
* Pregnancy
* History of major upper gastrointestinal surgery
* Allergy to ultrasound gel

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-05-19 (Actual); Study Completion 2024-05-26 (Actual)

PRIMARY OUTCOMES:
Gastric Residual Volume | before the study and 0, 10, 20, 30, 60, 90, 120 minutes after drinking the prepared drink each arm.If time to empty gastric antrum is extended, ultrasound will be serial performed at 150 and 180 minutes.
  gastric ultrasound at the gastric antrum by ultrasound

SECONDARY OUTCOMES:
Time to empty gastric antrum | 0, 10, 20, 30, 60, 90, 120 minutes after drinking the prepared drink each arm. If participants doesn't be empty stomach, time will extended to 120 and 180 minutes.
  Duration after drinking the drink until the gastric antrum cross-sectional area < 1.5 ml/kg measure by ultrasound
Point-of-care testing(POCT) glucose | Point-of-care testing(POCT) glucose is measured before the study, 60 and 120 after drinking the prepared drink each arm.
  measured by point-of-care testing(POCT) glucose at every 60 minutes entire the study
Hunger Numeric Rating Scale(NRS) | before the study, 60, and 120 minutes after drinking the prepared drink each arm
  Hunger will be measured by a numeric rating scale(NRS) before drinking, 60, and 120 minutes after drinking. The Numeric Rating Scale(NRS) is used for the self-report measurement of hunger levels, defined by numbers from 0 to 10, where 0 represents the lowest level of hunger and 10 represents the highest.
Thirst Numeric Rating Scale(NRS) | before the study, 60, and 120 minutes after drinking the prepared drink each arm
  Thirst will be measured by a numeric rating scale(NRS) before drinking, 60, and 120 minutes after drinking. The Numeric Rating Scale(NRS) is used for the self-report measurement of thirst levels, defined by numbers from 0 to 10, where 0 represents the lowest level of thirst and 10 represents the highest.
Nausea Numeric Rating Scale(NRS) | before the study, 60, and 120 minutes after drinking the prepared drink each arm
  Nausea will be measured by a numeric rating scale(NRS) before drinking, 60, and 120 minutes after drinking. The Numeric Rating Scale(NRS) is used for the self-report measurement of nausea levels, defined by numbers from 0 to 10, where 0 represents the lowest level of nausea and 10 represents the highest.

CONTACTS AND LOCATIONS:
Overall Officials: Chanya Deekiatphaiboon, Principal Investigator — Prince of Songkla University
Locations (1):
- Faculty of medicine, Songklanagarind Hospital, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No